CLINICAL TRIAL: NCT00974766
Title: Randomized Controlled Trial on the Efficacy and Safety of Two Different Glucocorticoid Dose Regimens in Allergic Bronchopulmonary Aspergillosis
Brief Title: Trial on the Efficacy and Safety of Two Different Glucocorticoid Dose Regimens in Allergic Bronchopulmonary Aspergillosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS/723/Res/276
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: bronchial asthma; allergic bronchopulmonary aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary; Asthma | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose glucocorticoid (Active Comparator): Low-dose steroid
  Interventions: Drug: Glucocorticoids
- High-dose glucocorticoid (Active Comparator): High-dose steroid
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Glucocorticoids — Prednisolone 0.5 mg/kg/day for 2 weeks; then 0.5 mg/kg/day for alternate days for eight weeks. Then taper by 5 mg every 2 weeks and discontinue
  Arms: Low-dose glucocorticoid
Drug: Glucocorticoids — Prednisolone 0.75 mg/kg/day for 6 weeks; then 0.5 mg/kg/day for 6 weeks. Then taper by 5 mg every 6 weeks and discontinue
  Arms: High-dose glucocorticoid

SUMMARY:
Allergic bronchopulmonary aspergillosis (ABPA) is a pulmonary disorder caused by a complex hypersensitivity response to antigens released by the fungus Aspergillus fumigatus. Oral corticosteroids are currently the treatment of choice for ABPA associated with bronchial asthma. They not only suppress the immune hyperfunction but are also anti-inflammatory. However, there is no data to guide the dose and duration of glucocorticoids and different regimens of glucocorticoids have been used in literature. The disorder is highly prevalent in India. The investigators have previously reported their experience with screening stable outpatients with bronchial asthma and acute severe asthma for ABPA. The investigators have also recently reported the prognostic factors associated with clinical outcomes in patients with ABPA.

The aim of this prospective randomized controlled trial (RCT) is to evaluate the efficacy and safety of two different glucocorticoid dose protocols in patients with ABPA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ABPA
* Presence of all the following three criteria:

  1. immediate cutaneous hyperreactivity on aspergillus skin test
  2. elevated total IgE levels > 1000 IU/mL
  3. A fumigatus specific IgE levels > 0.35 kU/L, AND,
* Presence of two of the following criteria:

  1. presence of serum precipitating antibodies against A fumigatus
  2. fixed or transient radiographic pulmonary opacities
  3. absolute eosinophil count > 1000/µL
  4. central bronchiectasis on HRCT

Exclusion Criteria:

* If they have taken glucocorticoids for more than three weeks in the preceding six months
* Failure to give informed consent
* Enrollment in another trial of ABPA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Glucocorticoid-dependent ABPA | two year
relapse rates in the two groups | one year

SECONDARY OUTCOMES:
time to first relapse | one year
glucocorticoid related adverse effects in the two groups | two years
response rates in the two groups | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, MD, DM, Principal Investigator — Postgraduate Institute of Medical Education and Research, Chandigarh, India
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Agarwal R, Aggarwal AN, Dhooria S, Singh Sehgal I, Garg M, Saikia B, Behera D, Chakrabarti A. A randomised trial of glucocorticoids in acute-stage allergic bronchopulmonary aspergillosis complicating asthma. Eur Respir J. 2016 Feb;47(2):490-8. doi: 10.1183/13993003.01475-2015. Epub 2015 Nov 19. PMID 26585431